CLINICAL TRIAL: NCT05550467
Title: 24-hour Urinary Electrolyte Excretion and Renal Prognosis in Chronic Kidney Disease：a Retrospective Cohort Study
Brief Title: 24-hour Urinary Electrolyte Excretion in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, LIANG Shuang, Dr., Chinese PLA General Hospital
Other Study IDs: 2015BAI12B06-03
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Diseases; Electrolyte Imbalance
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Association between excretion pattern and development trajectory of urinary electrolytes (urine sodium, urine potassium, urine chlorine, urine magnesium, urine calcium, urine phosphorus, urine creatinine, urea, uric acid, urine glucose, urine protein, urine retinol) and adverse prognosis in patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* Our study is a retrospective cohort study. The study included patients with adult（Age≥18years）CKD who were hospitalized in the Department of Nephrology, First Medical Center of Chinese PLA General Hospital from January 2014 to July 2022. Patients with CKD who had one or more 24-hour urinary electrolyte excretion tests at intervals of more than three months were included in the subgroup analysis.

Exclusion Criteria:

* Patients with hemodialysis therapy and urine volume less than 500ml were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years, chronic kidney disease patients without kidney replacement therapy who had 24-h urine eletrocyte tests.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Kidney disease progression | 2014.1.1-2022.7.31
  eGFR decline > 50%; dialysis; kidney transplant
Death | 2014.1.1-2022.7.31
  All cause death

SECONDARY OUTCOMES:
Cardiovascular disease | 2014.1.1-2022.7.31
  myocardial infarction, angina pectoris, stable heart failure, peripheral artery disease , revascularization, cerebrovascular events

IPD SHARING:
Plan to Share IPD: Undecided